CLINICAL TRIAL: NCT07139210
Title: EFFECT OF PERCEPTUAL-MOTOR TRAINING ON COGNITIVE FUNCTIONS, MOTOR ABILITIES AND QUALITY OF LIFE IN CHILDREN WITH ATTENTION DEFICIT HYPERACTIVE DISORDER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatalah khodair kamal abd_el_mageid, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012/005491
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Function; Quality of Life; ADHD - Attention Deficit Disorder With Hyperactivity; Motor Abilities
Keywords: PERCEPTUAL-MOTOR TRAINING; COGNITIVE FUNCTIONS; MOTOR ABILITIES; QUALITY OF LIFE; ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be assigned randomly into two groups of equal number . the randomization will be performed by sealed envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group A (No Intervention): Children in group A (control group) receive no treatment.
- experimental group B (Experimental): Children in group B (study group) are receiving the perceptual motor training program. Treatment program is applied for 60 minutes three days per week for three successive months.
  Interventions: Other: perceptual motor training

INTERVENTIONS:
Other: perceptual motor training — Perceptual -motor training program:
  1. Balance exercises
  2. Awareness training exercises
  3. Spatial awareness exercises
  4. Training of shape perception exercises
  5. Visual perception training exercises
  6. Auditory perception training
  7. Touch-kinetic perception training
  8. Coordination of eye and hand, eye and leg, subtle motor actions
  Arms: experimental group B

SUMMARY:
This study aims to Determine the effect of perceptual-motor training on:

cognitive functions, motor abilities, and quality of life in ADHD children.

DETAILED DESCRIPTION:
Thirty children with ADHD from both sexes are enrolled in this study. The selected children are randomly assigned by sealed envelopes into two groups of equal number 15 children for each group. Children in group A (control group) are receiving no treatment. Children in group B (study group) are receiving the perceptual motor training program. Treatment program is applied for 60 minutes three days per week for three successive months. All children will be assessed before and after the treatment program.

ELIGIBILITY:
Inclusion Criteria:

Age ranged from 8-12 years. Conner's score equal to or more than 65 according to hyperactivity index of conner's rating scale. Able to understand and follow instructions.

Exclusion Criteria:

Surgical interference in lower limbs and/or spine. Musculoskeletal problems or fixed deformities in the spine and/or lower extremities. Cardiovascular or respiratory disorders. Visual or hearing impairment. Receiving medical drugs that can cause confusion or make child less alert.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
cognitive functions: | 3 month
  Wechsler Intelligence Scale for Children-Fourth Edition (WISC-IV) is individually administered, and has 15 subtests. Each subtest is allocated to either the Verbal Comprehension (VC), Perceptive reasoning (PR), Working memory (WM), or Processing Speed (PS) subscales. The Full-scale IQ is composed of 10 core subtests: three VC (Vocabulary, Similarities, and Comprehension), three PR (Block Design, Picture Concepts, and Matrix Reasoning), two WM (Digit Span and Letter-Number Sequencing), and two PS (Coding and Symbol Search).
  As the scoring number increases it means a better outcome.

SECONDARY OUTCOMES:
motor ability | 3 month
  The Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) is used to assess following domains including Body co-ordination which consists of the following subtests: bilateral co-ordination. Balance. and strength and agility which consists of: running speed and agility subtest. Strength subtest.
quality of daily life | 3 month
  Pediatric Quality of Life Inventory Version 4.0 (PedsQL) is used for assessing quality of life as it's a multidimensional child self-report and parent proxy-report scales. It includes twenty-three items designed to measure dimensions of physical and psychosocial health as delineated by the world health organization.
  As scoring increases it means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Elsayed Shoukry, professor, Study Director — faculty of physical therapy
Locations (1):
- Faculty of Physical Therapy, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
could be not available